CLINICAL TRIAL: NCT00188539
Title: Predictive Assays in Cervix Cancer: Assessment of Hypoxia, Interstitial Fluid Pressure, and GSH Levels
Brief Title: Cervix:Hypoxia, Interstitial Fluid Pressure and GSH Levels
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Trials Group (Network); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 01-0376-C; National Cancer Inst of Canada
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cervix Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pre-treatment tumour oxygen measurements (under anesthesia) (Experimental)
  Interventions: Procedure: Pre-treatment tumour oxygen measurements (under anesthesia)

INTERVENTIONS:
Procedure: Pre-treatment tumour oxygen measurements (under anesthesia)

SUMMARY:
The aim of this study is to measure the oxygen content and interstitial fluid pressure in cervix cancer patients. Tumour oxygen content and internal pressure of tumours may be an important factor that influences the effectiveness of radiotherapy and other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with carcinoma of the cervix ( 3 cm in size or larger) where an examination under anesthesia is to be performed for staging purposes
* Informed consent

Exclusion Criteria:

* Patients with clinically occult cervix carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1995-12; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To determine if tumour oxygen tension prior to and during radiation therapy is an independent prognostic factor for primary tumour response and control in patients with cervix cancer. | tumour measurement will be done 2-3 months following completion of treatment; follow-up every 3 months for 2 years; every 4-6 months during year 3 to 5; and annually thereafter
To correlate tumour IFP measured before and during radiation therapy with oxygen tension as measured by the Eppendorf probe and to assess IFP as a prognostic factor for pelvic control. | tumour measurement will be done 2-3 months following completion of treatment; follow-up every 3 months for 2 years; every 4-6 months during year 3 to 5; and annually thereafter

SECONDARY OUTCOMES:
To determine if whole cell or nuclear GSH levels are correlated with tumour oxygen tension and with tumour response and control. | follow-up every 3 months for 2 years; every 4-6 months during year 3 to 5; and annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fyles, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada